CLINICAL TRIAL: NCT06739148
Title: The Enhancement Effect of Low-Level Laser Therapy for Muscle Training with Combined Neuromuscular Electrical Stimulation and Blood Flow Restriction
Brief Title: The Enhancement Effect of Low-Level Laser Therapy for Muscle Training with Combined NMES and BFR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-ER-113-089
Record Dates: First submitted 2024-09-12; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-09

CONDITIONS: Blood Flow Restriction Therapy; Neuromuscular Electrical Stimulation (NMES); Laser Therapy, Low-Level; Muscle Strength
Keywords: Muscle strength; Training; Low-level laser Therapy; Blood flow restriction; Neuromuscular electrical stimulation
MeSH Terms: interventions — Low-Level Light Therapy; Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LLLT+BFR+NMES (Experimental): LLLT: low-level laser therapy BFR: blood flow restriction NMES:neuromuscular Electrical Stimulation
  35 min/time, 3 times/weeks, 3 weeks
  Interventions: Device: Low Level Laser Therapy; Device: blood flow restriction; Device: Neuromuscular Electrical Stimulation
- BFR+NMES (Experimental): BFR: blood flow restriction NMES:Neuromuscular Electrical Stimulation
  35 min/time, 3 times/weeks, 3 weeks
  Interventions: Device: blood flow restriction; Device: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Device: Low Level Laser Therapy — Low-level laser therapy can increase cellular energy production, making it useful as a pre-conditioning treatment to prevent muscle contraction fatigue or as a post-contraction therapy to accelerate fatigue recovery.
  Arms: LLLT+BFR+NMES
Device: blood flow restriction — Its advantage is that during training, it can surpass the "overload principle," allowing for effective muscle cross-sectional area growth with relatively light weight training (20%-50% of 1RM or 20%-40% of MVC).
Device: Neuromuscular Electrical Stimulation — It is a strength training method that uses electrical currents to stimulate nerve and muscle activation, helping to maintain muscle mass, increase blood flow, and slow down or prevent muscle atrophy.

SUMMARY:
Blood flow restriction training (BFR) with neuromuscular stimulation (NMES) is employed for individuals with limited mobility and joint issues. However, this approach is highly susceptible to muscle fatigue, despite its potential beneficial effects on muscle strength. Recently, there has been growing interest in using low-level laser therapy (LLLT) to address muscle fatigue. LLLT, known for improving microcirculation and mitochondrial function, shows promise in alleviating enhanced muscle fatigue associated with combined BFR and NMES training. Despite these positive effects, there is limited knowledge about the short-term training impact of combined BFR and NMES with LLLT preconditioning. This project aims to investigate whether the photobiomodulation effects of LLLT could further enhance the training benefits of combined BFR and NMES. The study will employ an integrated analysis of decomposition surface EMG, EEG, and mechanomyogram to explore the behavior and neuromuscular mechanisms underlying the training benefits. If additional benefits are identified, LLLT pre-conditioning is recommended to enhance the use of combined BFR and NMES.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 20-40, without a diagnosis of cardiovascular or neuromusculoskeletal diseases.
2. Normal vision range after visual correction.

Exclusion Criteria:

1. Exclude students who have a teacher-student relationship with the principal investigator to ensure the participants' autonomy.
2. History of brain injury, stroke, spinal cord injury, or other neuromuscular-related conditions.
3. Contraindications for laser therapy: pregnancy, malignant tumor tissues, bleeding areas, and photosensitive skin regions.
4. Presence of any contraindications for blood flow restriction training, such as a history of injury or strain in the non-dominant arm's biceps, deep vein thrombosis or venous occlusion in the non-dominant arm, acute unstable fractures in the non-dominant arm, acute regional infections in the non-dominant arm, severe peripheral arterial occlusive disease in the non-dominant arm, complete lymphatic obstruction in the non-dominant arm, and edema due to acute pulmonary edema or congestive heart failure in the non-dominant arm.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Myoton | before training, 1week of training, 2 weeks of training, at the end of 3 weeks training
  Non-dominant hand extensor digitorum muscle belly parameters of static mechanical properties of muscles (Tone, Stiffness, Relaxation, Creep, etc.)
Mechanomyogram | before training, 1week of training, 2 weeks of training, at the end of 3 weeks training
  Recording of extensor digitorum muscle microshock waves during contraction
Multi-electrode surface EMG | before training, at the end of 3 weeks training
  Record muscle activity during contraction
Dynamometer System | before training, 1week of training, 2 weeks of training, at the end of 3 weeks training
  Measurement to track the degree of force applied by a non-dominant hand.

CONTACTS AND LOCATIONS:
Overall Officials: Ing-Shiou Hwang, PhD, Study Chair — NCKU, Institute of Allied Health Sciences
Locations (1):
- National Chen Kong University Hospital, Tainan, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No